CLINICAL TRIAL: NCT00479193
Title: Prospective Randomized Trial of Polymem vs. Bacitracin/Xeroform for Superficial Second Degree Burns
Brief Title: Polymem vs. Bacitracin/Xeroform in Treating Burn Wounds
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Charles J. Yowler MD, Doctor of Trauma Burns Surgery, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Investigator Initiated Trial
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Burns
Keywords: Burns; Dressing change
MeSH Terms: conditions — Burns | interventions — Bacitracin; 2,4,6-tribromophenol; Polymem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): There is one arm to the study. The same subjects are their own control. One of the investigators will identify two sites that appear to be the same depth on each patient [1 site Polymen and 1 site bacitracin/xeroform )]. One site will be identified for bacitracin/xeroform and one site for Polymen. All burns will be initially debrided and cleaned according to burn unit protocol. Laser Doppler will be utilized to determine burn depth at both the trial and control sites. On each subsequent visit, patients will rate the pain of the dressing change on a 1-10 pain intensity scale.The study will end for each patient when the investigator determines that 95% of their burn has re-epithelized.
  Interventions: Drug: bacitracin/xeroform; Drug: Polymem

INTERVENTIONS:
Drug: bacitracin/xeroform — single layer, change every 3 days
Drug: Polymem — single layer of Polymen, change every 3 days
  Other Names: No other names

SUMMARY:
Patients will be screened at the initial visit to the burn center. If the patients are eligible according to the inclusion/exclusion criteria, consent for the study will be obtained. One of the investigators will identify two sites that appear to be the same depth on each patient [1 site Polymen and 1 site bacitracin/xeroform )]. The depth of injury will be verified as partial thickness using laser doppler. Each site will be at least 4cm x 4cm in size. One site will be identified for bacitracin/xeroform and one site for Polymen. All burns will be initially debrided and cleaned according to burn unit protocol. The dressing will then be applied. All dressings will be covered with cotton gauze and ace wraps. Laser Doppler will be utilized to determine burn depth at both the trial and control sites. On each subsequent visit, patients will rate the pain of the dressing change on a 1-10 pain intensity scale. It will be noted if the wound appears infected or if antibiotics are prescribed.

The study will end for each patient when the investigator determines that 95% of their burn has re-epithelized.

DETAILED DESCRIPTION:
Superficial second degree burns are limited to the epidermis and superficial layer of the dermis and are expected to heal without the need of surgery if they are treated appropriately. Complications such as desiccation of the wound or infection may extend the depth of the injury and result in an increase in scarring or the requirement for excision of the burn and skin grafting. The MetroHealth Burn Center treats over 1500 patients a year for superficial second degree burns.

Various methods are used from the conventional dressing methods using guaze to the methods that use biological materials such as skin from cadavers, pig's skin and artificial synthetic materials. Our present burn care involves initial superficial outpatient debridement of the burn wound and application of a dressing. This dressing consists of bacitracin applied to the burn wound and xeroform covered by cotton gauze and ace-wrap. The majority of our patients are unable to change this dressing by themselves and they either return to the burn center daily for wound care or we arrange for a visiting nurse.

Polymem is a novel dressing which has been approved by the FDA for open wounds including burns.Polymem is a hydrophilic polyurethane membrane pad with a semi permeable polyurethane film backing. The pad contains a wound cleanser (F68 surfactant), a moisturizer (glycerin) and an absorb ing agent (super-absorbent polymem). The F86 surfactant is involved in dissolving the superficial necrotic layer of the burn and helps clean the burn site. Glycerin acts as a moisturizer and prevents the pad from sticking to the wound. The absorbing agent maintains the moisture of the wound which has been shown to increase wound healing. It also allows the dressing to remain on the wound for three days. Kim et al conducted a study of 44 patients with second degree burns and demonstrated an increase in healing time, more comfort, and a decrease in dressing changes with the use of Polymem.

ELIGIBILITY:
Inclusion Criteria:

1. Age + to or greater than 18
2. Superficial 2nd degree burns of the trunk and extremities which the evaluating investigator believes will heal within 21 days without the need for surgery.
3. Burn injury is less than 48 hours old
4. Patient is able to return to burn clinic for required follow-up.
5. Burn is of sufficient size to permit the application of trial and control dressings
6. Outpatient

Exclusion Criteria:

1. Age under 18
2. Burn injury over 48 hours old
3. Deep burn not expected to heal within 21 days
4. Extremely superficial burn expected to heal in less than 7 days.
5. Infected burns
6. Patient unable to return to clinic for required follow-up (i.e. will use visiting nurse or PCP for follow-up).
7. Patient unable to give consent.
8. Inpatient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10 (Estimated); Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Time to wound healing | 21 days

SECONDARY OUTCOMES:
Comparing two FDA cleared products for decreased frequency of dressing changes to every third day, less pain, decrease in infection, and cost effectiveness. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Yowler, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Carr RD, Lalagos DE. Clinical evaluation of a polymeric membrane dressing in the treatment of pressure ulcers. Decubitus. 1990 Aug;3(3):38-42. PMID 2205233
- [Background] Agren MS, Mertz PM, Franzen L. A comparative study of three occlusive dressings in the treatment of full-thickness wounds in pigs. J Am Acad Dermatol. 1997 Jan;36(1):53-8. doi: 10.1016/s0190-9622(97)70325-6. PMID 8996261
- [Background] Fowler E, Papen JC. Clinical evaluation of a polymeric membrane dressing in the treatment of dermal ulcers. Ostomy Wound Manage. 1991 Jul-Aug;35:35-8, 40-4. No abstract available. PMID 1878118
- [Background] Blackman JD, Senseng D, Quinn L, Mazzone T. Clinical evaluation of a semipermeable polymeric membrane dressing for the treatment of chronic diabetic foot ulcers. Diabetes Care. 1994 Apr;17(4):322-5. doi: 10.2337/diacare.17.4.322. PMID 8026290